CLINICAL TRIAL: NCT01660724
Title: Ultrasound Guided Arterial Puncture: a Prospective, Blinded, Randomised Controlled Trial.
Brief Title: Ultrasound Guided Arterial Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Christian Borbjerg Laursen, Principal investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Mulvarp2012
Record Dates: First submitted 2012-07-16; First posted 2012-08-09 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Arterial Puncture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided arterial puncture (Experimental): Patients randomised to the this arm has arterial puncture performed using simultaneously ultrasound in order to guide the passage of the syringe from the patient's skin to the artery
  Interventions: Procedure: Ultrasound guided arterial puncture
- Conventional arterial puncture technique (Active Comparator): Patients randomised to the active comparator arm has arterial puncture performed using the conventional technique
  Interventions: Procedure: Conventional arterial puncture technique

INTERVENTIONS:
Procedure: Ultrasound guided arterial puncture — Arterial puncture is performed using simultaneously ultrasound in order to guide the passage of the syringe from the patient's skin to the artery
  Arms: Ultrasound guided arterial puncture
Procedure: Conventional arterial puncture technique — Arterial puncture is performed using the conventional technique
  Arms: Conventional arterial puncture technique

SUMMARY:
The main purpose of the study is to evaluate whether the routine use of ultrasound guided arterial puncture can increase the proportion of patients who only needs one puncture attempt in order to successfully extract enough blood to make an arterial blood gas analysis, when ultrasound guided arterial puncture is compared to conventional arterial puncture technique.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted or treated in the acute emergency department
* Indication for a arterial blood gas analysis, according to the physician responsible for the patient's hospital stay / treatment

Exclusion Criteria:

* Patient age < 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2012-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who only needs one puncture attempt in order to successfully extract enough blood to make an arterial blood gas analysis | up to 1 hour after arterial puncture

SECONDARY OUTCOMES:
Time used for arterial puncture | up to 1 hour after arterial puncture
Patient corporation | up to 1 hour after arterial puncture
  Patient corporation is subjectively estimated by the physician performing the arterial puncture. The degree of patient corporation are assessed on a scale from 1 - 5, where 1 is very poor patient corporation and 5 is perfect patient corporation.
Pain Scores on the Visual Analog Scale | Up to 1 hour after arterial puncture
Number of attempts before successfully acquiring arterial puncture | up to 1 hour after arterial puncture

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Laursen, MD, Principal Investigator — Odense Universityhospital
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140